CLINICAL TRIAL: NCT06110767
Title: The Effects of a Healthy Nutrition Program and Virtual Reality Applications on Body Composition and Physical Fitness in Female Individuals.
Brief Title: The Effects of a Healthy Nutrition Program and Virtual Reality Applications on Body Composition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erzurum Technical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bozkurt.osman
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Obesity; Virtual Reality; Body Composition; Healthy Nutrition; Physical Fitness
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: This research is a cross-sectional, prospective and experimental study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Routine diet + Non-immersive virtual reality-based physical activity application (Experimental): Non-immersive virtual reality will be applied 30 minutes a day, 3 days a week for 4 weeks.
  Interventions: Device: non-immersive virtual reality
- Diet Program for healthy eating + Non-immersive virtual reality-based physical activity app (Experimental): In addition to the 4-week diet program,Non-immersive virtual reality will be applied 30 minutes a day, 3 days a week for 4 weeks.
  Interventions: Device: non-immersive virtual reality; Behavioral: Healty Diet Programme
- Diet program for healthy eating (Experimental): 4-week diet program will be applied.
  Interventions: Behavioral: Healty Diet Programme

INTERVENTIONS:
Device: non-immersive virtual reality — Non-Immersive Virtual Reality Based Physical Activity Application: Application will be carried out 3 days a week, 30 minutes a day, for 4 weeks. Kinect Adventures and Kinect Sports game packages will be used using the Microsoft Kinect Xbox 360 game console. It is planned that the participants will engage in physical activity with these game packages.
  Arms: Diet Program for healthy eating + Non-immersive virtual reality-based physical activity app; Routine diet + Non-immersive virtual reality-based physical activity application
Behavioral: Healty Diet Programme — Healthy nutrition program: It will be implemented for 4 weeks.Healthy Nutrition Program: Türkiye Ministry of Health nutrition program will be prepared based on the recommendations of the Turkey Nutrition Guide published by the Ministry of Health in 2016 (TÜBER-2016). A personalized healthy nutrition program will be created in line with this guide, taking into account the age, gender and physical activity status of healthy individuals.
  Arms: Diet Program for healthy eating + Non-immersive virtual reality-based physical activity app; Diet program for healthy eating

SUMMARY:
The most commonly used method in the management of body compositions of healthy individuals in the recent times is the application of physical activity together with a healthy nutrition (diet). The application of diet together with physical activity cause significant changes in the body composition (fat ratio, muscle mass, lean body mass, etc.). Physical activity can be done with traditional physical activity methods as well as with virtual reality applications. Virtual reality is a simulation or a metaversal facet of a real environment created by a computer or various other electronic devices that allows one or more users to interact with certain elements in a simulated virtual frame through a human-machine interface. Virtual reality applications are generally classified as immersive and non-immersive virtual reality . Commercial games such as Sony Playstation, Microsoft Kinect Xbox 360, Nintendo Wii can be given as examples of non-immersive virtual reality . In order to preserve body composition, different exercise applications can be recommended in addition to the diet program. In the literature, many studies involving diet, physical activity or a combination of these two applications have been experimentally planned and carried out in a controlled manner. In these studies, moderate body weight loss (1-5 kg) was reported with only physical activity. It is a general opinion that diet therapy in addition to planned physical activity (exercise) provides more effective and healthier results than people who lose weight with only diet programs or only exercise. It has been stated in previous studies that body composition and physical fitness improve with virtual reality application as happened wih diet intervention. However, due to the fact that access to virtual reality applications is not very easy, longitudinal studies are needed to evaluate whether they should be included in general body composition and physical fitness improvement programs. At this point, the main purpose of this study is to compare and evaluate the effects of virtual reality applications and healthy nutrition program on improving body composition and physical fitness.

DETAILED DESCRIPTION:
Physical inactivity is one of the main causes of many diseases. The development of technology causes some activities in daily life not to be performed and physical activity to decrease. Many diseases such as obesity, cardiovascular diseases and diabetes are more common in inactive and sedentary individuals.

In order to maintain body weight in sedentary individuals, the energy intake and expenditure must be equal. Today, mechanized social life reduces physical activity and keeps the energy that needs to be spent in the body, and this accumulation negatively affects the balance of energy intake and expenditure. In recent years, the increased consumption of highly processed food and beverages has caused changes in the world's diet. The main changes observed include imbalance in energy intake, change in eating frequency, and faster production and consumption of food. Obesity is not only among adults due to the decrease in physical activity in the world and in our country, the time spent in front of the television and computer reaching serious levels, high-energy - high-fat foods becoming more accessible and cheaper, and the rapid increase in industrial food production that is rich in salt but poor in fiber and vitamins; It is also seen among children and adolescents.

The most commonly used method today in the management of body composition of healthy individuals is the implementation of physical activity along with healthy nutrition (diet). Application of diet along with physical activity creates significant changes in body composition (fat ratio, muscle mass, lean body mass, etc.). Physical activity can be done with traditional physical activity methods or with virtual reality applications.

Virtual reality is a simulation or metaversal aspect of a real environment created by a computer or other various electronic devices that allows one or more users to interact with certain elements in a simulated virtual framework through a human-machine interface. Virtual reality applications are generally classified as immersive and non-immersive virtual reality . In immersive virtual reality, the user's interaction with the real world is usually limited by using virtual reality glasses. In non-immersive virtual reality, the user can manipulate the avatars on the screen, thanks to sensors that detect body movements, in order to maintain their connection with the outside world. Non-immersive virtual reality applications generally include a display, a receiving sensor, and a main application device. Commercial games such as Sony Playstation, Microsoft Kinect Xbox 360, Nintendo Wii can be given as examples of non-immersive virtual reality.

It has been observed that the use of virtual reality applications as a rehabilitation approach in various diseases has increased over the last 2 decades. It is seen to be used in areas such as stroke rehabilitation, various psychotherapy applications, improving physical fitness and improving body composition. Physical activity and nutrition are one of the few consistent factors associated with body composition. In addition to the diet program, different exercise practices can be recommended to maintain body weight. In the literature, many studies involving diet, physical activity, or combinations of these two practices have been experimentally planned and carried out in a controlled manner. In these studies, moderate body weight losses (1-5 kg) were reported only with physical activity . It is a general opinion that a healthy nutrition program, in addition to planned physical activity (exercise), provides more effective and healthy results than people who lose weight with diet programs or exercise alone. Just as body composition and physical fitness improve thanks to diet practices, it has been stated in previous studies that changes in body composition are also observed thanks to virtual reality-based physical activity applications. However, since access to virtual reality applications is not very easy, longitudinal studies are needed to evaluate whether they should be included in programs to improve general body composition and physical fitness.

The aim of this study is to compare and evaluate the effects of virtual reality-based physical activity applications and a healthy nutrition program on improving body composition and physical fitness.

The sample of the study will be female adult volunteers. The total number of participants required for the study to provide 92% accuracy was calculated as 27 people in the G power 3.1 program, based on the study of Zeng et al. (2021). A consent form will be obtained from each participant. Approval was received for this research from Erzurum Technical University Ethics Committee.

The sample of the study will consist of healthy individuals between the ages of 18-64 who do not have any health problems and do not need a special diet, living in Erzurum.

Exclusion criteria of the study: BMI value of 40.0 and above will prevent the implementation of a healthy nutrition program and virtual reality-based physical activity applications.

having situations. A total of 45 healthy individuals are planned to participate in the study. Participants will be classified into three groups using the stratified randomization method so that their current Body Mass Index (BMI) average and physical activity levels are equal. There will be 15 participants in each group.

ELIGIBILITY:
Inclusion Criteria:

* Having BMI value between 25.0-39.9
* Female gender
* Volunteer between the ages of 18-64
* Not having any cardiovascular or orthopedic problems that would prevent attendance

Exclusion Criteria:

* Having a BMI value of 40.0 and above
* Having conditions that would prevent the implementation of a healthy nutrition program and virtual reality-based physical activity practices.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — It will consist of healthy female individuals between the ages of 18-64.
Enrollment: 45 (Estimated)
Dates: Start 2023-11-20 (Estimated); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Body composition | Change from baseline body composition at week 4
  The height of the participants will be determined with the Tanita Stadiometer with an accuracy of 0.01 mm. Body weights, Body Mass Index (BMI), Body fat percentage, Total fat mass, muscle mass, bone mass, etc. A lot of data regarding body composition will be recorded using the Tanita body analyzer. Individuals' height and body analysis will be carried out in accordance with measurement techniques.
Waist to hip ratio | Change from baseline waist to hip ratio at week 4
  It will be carried out with a non-flexible tape measure and the waist and hip values will be proportional to each other.
Functional Capacity | Change from baseline functional capacity at week 4
  6-minute walk test: In the 6-minute walk test, the patient walks as fast as he can in a straight corridor of at least 30 meters, but without running. It is measured how many meters he walked. The patient should not change his tempo and speed during the test.
Balance | Change from baseline dynmic balance at week 4
  The Y Balance Test (YBT) is a simple, yet reliable, test used to measure dynamic balance.The YBT requires the athlete to balance on one leg whilst simultaneously reaching as far as possible with the other leg in three separate directions: anterior, posterolateral, and posteromedial. Therefore, this test measures the athlete's strength, stability and balance in various directions. The YBT composite score is calculated by summing the three reach directions and normalising the results to the lower limb length, whereas asymmetry is the difference between right and left limb reach (1) - this is explained in greater detail in the scoring system section.

SECONDARY OUTCOMES:
Dynamic Balance | Change from baseline dynmic balance at week 4
  Functional Reach Test (FRT) is a clinical outcome measure and assessment tool for ascertaining dynamic balance in one simple task.The patient is instructed to stand next to, but not touching, a wall and position the arm that is closer to the wall at 90 degrees of shoulder flexion with a closed fist.
  The assessor records the starting position at the 3rd metacarpal head on the yardstick.
  Instruct the patient to "Reach as far as you can forward without taking a step." The location of the 3rd metacarpal is recorded. Scores are determined by assessing the difference between the start and end position is the reach distance, usually measured in inches.

CONTACTS AND LOCATIONS:
Overall Officials: Betül KOCAADAM_BOZKURT, PhD, Study Director — Erzurum Technical University

IPD SHARING:
Plan to Share IPD: No